CLINICAL TRIAL: NCT06619613
Title: A Randomized, Double-blind, Placebo-controlled and Multiple Dose Escalation Phase Ib Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of CM383 in Patients With Alzheimer's Disease Related Mild Cognitive Impairment and Mild Alzheimer's Disease
Brief Title: A Study of CM383 in Patients With Alzheimer's Disease Related Mild Cognitive Impairment and Mild Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM383-109001
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Amyloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): CM383 injection, Intravenous infusion
  Interventions: Biological: Alzheimer Disease (AD); Other: Placebo
- Group 2 (Experimental): CM383 injection, Intravenous infusion
  Interventions: Biological: Alzheimer Disease (AD); Other: Placebo
- Group 3 (Experimental): CM383 injection, Intravenous infusion
  Interventions: Biological: Alzheimer Disease (AD); Other: Placebo
- Group 4 (Experimental): CM383 injection, Intravenous infusion
  Interventions: Biological: Alzheimer Disease (AD); Other: Placebo

INTERVENTIONS:
Biological: Alzheimer Disease (AD) — CM383 injection
Other: Placebo — Matched placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled and multiple dose escalation phase Ib study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of CM383 in patients with Alzheimer's disease related mild cognitive impairment and mild Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate and have the subject and their legal guardian jointly sign the Informed Consent Form.
* The age of the subjects is between 50 and 85 years old.
* BMI≥19kg/m2 and ≤32.5 kg/m2, weight ≥45 kg and ≤100 kg at screening or baseline.

Exclusion Criteria:

* Cognitive impairment of subjects due to other medical or neurological factors (other than AD)
* History of stroke or transient ischemic attack, seizures, or other unexplained loss of consciousness within the past year
* With any mental illness that may interfere with the cognitive assessment of the subjects.
* With history of moderate or severe renal dysfunction.
* With Uncontrolled stable hypertension.
* With history of severe trauma or major surgery in the 6 months prior to the screening period, or planned surgery during the study.
* History of malignancy within 5 years prior to screening.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse event | Up to Week 26
  The occurrence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Shi, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, China